CLINICAL TRIAL: NCT03699683
Title: A Supervised Exercise Program After Bariatric Surgery Avoids Fat-Free Mass Loss And Reduces Cardiovascular Risk Factors
Brief Title: Physical Activity Program After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Manuel Moya, Principal Investigator, Universidad Miguel Hernandez de Elche
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015.60.E.OEP
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Bariatric Surgery and Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: two groups (experimental and control) randomly assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Combined Activity Program (Experimental): Before and after a 6-months supervised and individualized program that combined aerobic and resistance training were performed in post bariatric patients. Body composition, physical fitness and cardiovascular risk factors were measured before, after the physical activity program and 6 months later (13 months sinde the program started)
  Interventions: Other: Combined aerobic and resistance training program

INTERVENTIONS:
Other: Combined aerobic and resistance training program

SUMMARY:
Background: Bariatric surgery (BS) causes large weight reductions and improvements in cardiovascular risk (CVR), although, there are also decreases in fat-free mass (FFM). However, the effects of exercise after surgery on these variables remains to be determined.

Methods: 38 patients who underwent BS were divided into two groups: an experimental group (EG, n = 19) and a control group (CG, n = 19). Body composition, physical fitness, CVR and CVR factors were assessed in both groups one month after the surgery (T1), at 7 months (T2) and at 13 months (T3). Between T1 and T2, the EG performed a 6 month monitored aerobic and resistance combined training.

DETAILED DESCRIPTION:
Forty adults that underwent BS (sleeve gastrectomy and gastric bypass) were invited to participate in the study along two years (between 1-4 patients per month). After the initial interview, two patients refused to participate in the study. The participants provided written informed consent before starting the study. The study was approved by the Ethics Committee of the University in accordance with the Declaration of Helsinki. Participants were divided into two groups (experimental, EG; and control, CG) depending on when the BS was performed. The first 10 patients of each year were the EG (n=19) and the other mine patients were the CG (n=19). A 6-month supervised and individualized program that combined aerobic and resistance training (CART) was only conducted with the EG. Both groups followed a nutritional supervision and were evaluated in 3 different time periods: Test 1 (T1), before the intervention period (approximately 1 month after BS) with no differences in any variable measured; Test 2 (T2), after the intervention period (7 months after BS) and Test 3 (T3) to evaluate a retention period (13 months after BS). The tests included in the evaluation were: blood sample, body composition, blood pressure, physical fitness (cardiorespiratory fitness, isokinetic and isometric strength measures of the lower limbs) and CVR. The test protocols were divided into 3 days: 1) between 8:00 AM and 9:00 AM., a blood sample was collected. 2) 24 hours after, at the same hour, body composition and resting blood pressure were measured. In the afternoon (between 5:00 P.M. and 8:00 P.M.), muscle strength measures were obtained. 3) at least 72 hours after the second testing session day, a cardiorespiratory fitness test was performed. Body composition, blood pressure and strength and cardiovascular tests were conducted at the facilities of the Sports Research Centre (Elche, Spain), in a climatically controlled laboratory, with a temperature between 22-24º and relative air humidity between 45-60%. Before any testing, all participants attended two familiarization sessions to introduce testing procedures and minimize the learning effects over the measures

ELIGIBILITY:
Inclusion Criteria:

1. Meet the age requirements
2. Be a patient of the reference hospital.
3. Follow the doctor's usual health prescriptions

Exclusion Criteria:

1. Cardiovascular diseases
2. Chronic respiratory deseases
3. Cancer in the 5 years prior to surgery
4. Severe functional limitations

Ages: 35 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (T1) Total Cholesterol Blood Samples at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  Blood samples were taken at the Vinalopó-Salud Hospital of Elche (Spain), after a 12 h fast and 48 h before the test and without performing exercise in that period. Total cholesterol was measured using standard methods.
Change from Baseline (T1) HDL Cholesterol Blood Samples at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  Blood samples were taken at the Vinalopó-Salud Hospital of Elche (Spain), after a 12 h fast and 48 h before the test and without performing exercise in that period. HDL cholesterol was measured using standard methods.
Change from Baseline (T1) Glucose Blood Samples at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  Blood samples were taken at the Vinalopó-Salud Hospital of Elche (Spain), after a 12 h fast and 48 h before the test and without performing exercise in that period. Glucose was measured using standard methods.
Change from Baseline (T1) Triglycerides Blood Samples at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  Blood samples were taken at the Vinalopó-Salud Hospital of Elche (Spain), after a 12 h fast and 48 h before the test and without performing exercise in that period. Triglycerides were measured using standard methods.
Change from Baseline (T1) Body composition at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  Body mass index (BMI) was calculated according to the formula: total weight in kilograms divided by squared height in meters (kg·m-2). Participants performed the assessment with an empty bladder. Bioimpedance analysis (Tanita, TBF 300A, Tokyo, Japan) was used to establish body weight and body composition.
Change from Baseline (T1) waist and hip circumference at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  The ISAK (International Society for the Advancement of Kinanthropometry) protocol was used to assess waist and hip circumference.
Change from Baseline (T1) Systolic and Diastolic Blood pressure at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  A digital sphygmomanometer (Microlife WatchBP Home, Heerbrugg, Switzerland) was used to measure blood pressure, according to established recommendations.
Change from Baseline (T1) Cardiorespiratory Fitness at 13 months | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 8:00 AM and 9:00 AM.
  The maximum oxygen consumption (VO2max) was determined indirectly following the protocol previously published (YMCA) on a cycle ergometer (Technogym Bike Med, Technogym, Gambettola, Italy). The VO2max was calculated using the following formula: VO2max (ml·Kg-1·min-1) = 1.8 *(6.12 * Wpeak) / BW + 3.5 + 3.5 (in which "BW" is body mass in kilograms and "Wpeak" is the power output in watts). Additionally, VO2max was expressed in absolute values (VO2max abs), relative to FFM (VO2max/FFM) and relative to each individual's body weight (VO2max/BW). A digital sphygmomanometer (Tango+, Suntech, USA) was used for the assessment of blood pressure and an electrocardiogram was also administered. An experienced exercise physiologist together with a cardiologist supervised all the cardiorespiratory tests.
Change from Baseline (T1) Muscle strength at 13 months. Range of Motion of Dynamic strength measurement | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 5:00 PM and 8:00 PM.
  Participants performed 1 submaximal trial (1st set) to get used to the range of motion and the accommodating resistance of the dynamometer.
Change from Baseline (T1) Muscle strength at 13 months. Dynamic strength measurement | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 5:00 PM and 8:00 PM.
  Participants performed 3 sets of 4 concentric contractions (flexion-extension) of lower body (knee), at an angular speed of 60º/s, with 90 s rest between repetitions. The knee motion ranges were within 105° to 10°. The participants were verbally encouraged to perform and maintain maximal effort in every contraction. The peak torque (N·m) of each set was analyzed and the average of the last three sets was calculated. Additionally, the peak torque was normalized to the individual's body weight (N·m·kg-1∙100) and relative to FFM (N·m·FFM-1∙100).
Change from Baseline (T1) Muscle strength at 13 months. Isometric strength measurement | Baseline (T1), at 7 months (T2) and at 13 months (T3), between 5:00 PM and 8:00 PM.
  Participants completed four repetitions of a Maximum Voluntary Contraction trial (15 s rest between repetitions), during which they were verbally encouraged to perform a maximal effort for 5 s. The first repetition was a submaximal familiarization trial. The angles used for assessing quadriceps and hamstrings were of 105º and 75º, respectively. As there was one set per exercise, the peak torque (N·m) was analyzed and normalized to each participant´s body weight (N·m·kg-1∙100) and individual FFM (N·m·FFM-1∙100).

IPD SHARING:
Plan to Share IPD: Undecided